CLINICAL TRIAL: NCT03791294
Title: Trial on the Use of Microcrystalline Titanium Dioxide With Covalently Linked Monovalent Silver Ions (TIAB) in the Formulation of Vaginal Capsules in the Prevention of Complications After Total Hysterectomy
Brief Title: Effects of Microcrystalline Titanium Dioxide With Covalently Linked Monovalent Silver Ions on Complications After Total Hysterectomy ( ISTIAB-0)
Acronym: ISTIAB-0
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Simone Garzon, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISTIAB-0
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Infection; Bleeding; Complication, Postoperative
MeSH Terms: conditions — Infections; Hemorrhage; Postoperative Complications | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIAB treatment (Experimental): From the first postoperative day for ten days, single vaginal capsule per day of TIAB (microcrystalline titanium dioxide with covalently linked monovalent silver ions), Sodium Hyaluronate, and Aloe Barbadensis Extract vaginal capsule.
  Interventions: Drug: TIAB: microcrystalline titanium dioxide with covalently linked monovalent silver ions
- Control (No Intervention): No treatment

INTERVENTIONS:
Drug: TIAB: microcrystalline titanium dioxide with covalently linked monovalent silver ions — TIAGIN vaginal capsule, composition: TIAB (microcrystalline titanium dioxide with covalently linked monovalent silver ions), Sodium Hyaluronate, Aloe Barbadensis Extract
  Other Names: TIAGIN vaginal capsule, composition: TIAB (microcrystalline titanium dioxide with covalently linked monovalent silver ions), Sodium Hyaluronate, Aloe Barbadensis Extract
  Arms: TIAB treatment

SUMMARY:
Total hysterectomy is one of the most performed surgical procedures in the world and it is associated with post-operative complications. The postoperative morbidity rate is estimated to vary from 3% to 8% with a readmission rate of 5-7%. The most frequent postoperative complications are urinary tract infections, wound infection of the vaginal vault, vault cellulitis, bleeding, suture dehiscence, pelvic abscess. The introduction of routine antibiotic prophylaxis has significantly reduced the risk of infectious complications, which however remains higher than other "clean" surgery, mainly due to contamination by the vaginal bacterial flora. In this scenario, the introduction of adjuvant factors acting on bacterial flora, can contribute to reduce the risk of post-surgical complications.

The cationic silver ions (Ag +) stabilized by covalent link with Titanium dioxide (TiO2), the TIAB, maximizes the properties of silver by optimizing the antibiotic action and disruptive properties of the pathogenic biofilm of bacteria and fungi. Thanks to these properties, TIAB is able to enhance the antibiotic action by reducing the risk of antibiotic resistance and recurrent infections linked to the biofilm. Re-establishing the optimal vaginal microenvironment represents a fundamental step reducing the risk of infections in the surgical site, since the vagina is a non-sterile environment populated by bacterial species that can generate biofilm and potentially infect the site of surgery. In addition to microbicidal and disruptive biofilm activity, TIAB has demonstrated a direct action on tissue regeneration processes by stimulating the production of collagen and its modeling.

Different clinical trials have reported a cicatrizing and re-epithelializing action of TIAB administered vaginally in the context of cervical conization for pathology related to HPV. Without showing any notable adverse effects or a negative action on lactobacillary flora with an overall good therapy tolerance by patients.

On the basis of the available evidence, the investigators conduct a randomized controlled clinical trial to determine if TIAB treatment in the formulation of vaginal capsules TIAGIN (TIAB (microcrystalline titanium dioxide with covalently linked monovalent silver ions), Sodium Hyaluronate, Aloe Barbadensis Extract) is able to reduce the incidence of infectious complications, that are related to altered healing of post-hysterectomy vaginal suture.

ELIGIBILITY:
Inclusion Criteria:

* Women underwent laparoscopic total hysterectomy for benign gynecological pathology

Exclusion Criteria:

* Women underwent non-laparoscopic total hysterectomy
* Women underwent laparoscopic total hysterectomy for malignant pathology
* Patients with diabetes mellitus in insulin therapy
* Smoking patients
* Patients suffering from chronic rheumatic diseases or chronic diseases not in adequate control.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal bleeding | At the 30th post operative day
  at least one episode of red vaginal blood loss
Vaginal vault infection | At the 30th post operative day
  at least one episode of inflammation and infection in the vaginal vault suture requiring antibiotic therapy
Urinary tract infection | At the 30th post operative day
  at least one episode of signs and symptoms requiring empiric antibiotic therapy
Dehiscence of vaginal vault suture | At the 30th post operative day
  Dehiscence of vaginal vault suture requiring repeat surgery
Readmission | At the 30th post operative day
  At least one episode of readmission related to postoperative complications

SECONDARY OUTCOMES:
Adverse events | At the 30th post operative day
  Adverse events due to the use of vaginal capsule therapy: erythema, vaginal and vulvar pruritus, dermatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Garzon, M.D., Principal Investigator — Università degli Studi dell'Insubria; Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Fabio Ghezzi, M.D., Principal Investigator — Università degli Studi dell'Insubria; Jvan Casarin, M.D., Principal Investigator — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided